CLINICAL TRIAL: NCT00003013
Title: European Cooperative Study of Chemotherapy and Surgery Comparing Adjuvant Doxorubicin Followed by CMF vs. Adjuvant Doxorubicin/Paclitaxel Followed by CMF vs. Primary Doxorubicin/Paclitaxel Followed by CMF in Women With Operable Breast Cancer and T>2 cm
Brief Title: Chemotherapy Plus Surgery in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065593; INT-23/96; EU-97001
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2000-06

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — CMF regimen; Cyclophosphamide; Doxorubicin; Fluorouracil; Methotrexate; Paclitaxel; Tamoxifen; Radiotherapy

INTERVENTIONS:
Drug: CMF regimen
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: fluorouracil
Drug: methotrexate
Drug: paclitaxel
Drug: tamoxifen citrate
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining surgery with chemotherapy may kill more tumor cells. It is not yet known which treatment regimen is more effective for breast cancer.

PURPOSE: Randomized phase III trial to study the effectiveness of chemotherapy plus surgery in treating women who have breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate whether 8 courses of primary chemotherapy before adequate surgery of breast tumor and locoregional radiotherapy plus tamoxifen for 5 years improves the disease-free and overall survival in women with operable breast carcinoma and tumor at diagnosis greater than 2 cm in diameter.
* Assess whether, in the postoperative arms, the addition of paclitaxel to doxorubicin before CMF (cyclophosphamide, methotrexate, and fluorouracil) improves disease-free and overall survival in these patients.
* Define the incidence of pathologic complete response (CR) induced by 8 courses of primary chemotherapy containing paclitaxel.
* Assess whether a pathologic CR is an independent predictor of disease-free and overall survival.
* Evaluate the effects of primary chemotherapy on the rate and quality of breast conserving surgery.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by center, tumor diameter at mammography, nuclear or histological grade, and estrogen/progesterone receptor status. Patients are randomized to one of three treatment arms.

* Arm I: Patients receive doxorubicin IV over 15 minutes once every 3 weeks for 4 courses. Beginning 21 days after the last administration of doxorubicin, patients receive cyclophosphamide IV, methotrexate IV, and fluorouracil IV on days 1 and 8. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
* Arms II and III: Patients receive doxorubicin IV over 15 minutes and paclitaxel IV over 3 hours once every 3 weeks for 4 courses. Beginning 21 days after the last administration of doxorubicin and paclitaxel, patients receive cyclophosphamide IV, methotrexate IV, and fluorouracil IV on days 1 and 8. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

All patients have either mastectomy or breast conserving surgery; patients with unclear surgical margins may have second surgery (re-resection or total mastectomy) or radiotherapy. Lymph node axillary dissection is performed up to at least the second level. For patients in the 2 adjuvant arms (arms I and II), adjuvant chemotherapy starts by day 21 after surgery. For patients in the primary chemotherapy arm (arm III), surgery is performed by day 28 after the last course of chemotherapy or at resolution of all possible hematological or infective complications.

At the end of the combined surgery plus chemotherapy approach (i.e., after the last course of CMF (arms I and II) or after surgery (arm III)), patients enrolled after June 30, 2000 with estrogen or progesterone receptor positive disease receive oral tamoxifen daily for 5 years.

All patients who have breast conserving surgery receive postoperative irradiation within 4 weeks after completing chemotherapy and surgery (i.e., within 4 weeks from last dose of adjuvant chemotherapy (arms I and II) or from surgery (arm III)). All patients who have mastectomy and have pT4 disease must receive irradiation to the chest wall.

Patients are followed at 6, 12, 18, and 24 months, and then annually thereafter.

PROJECTED ACCRUAL: A total of 450 patients per arm will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Unilateral carcinoma of the breast that has not been previously treated with standard therapies
* Tumor greater than 2 cm in its maximum diameter as assessed by mammography, except:

  * No locally advanced disease, i.e., no tumor with direct extension to the chest wall or skin
  * No metastatic disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Karnofsky 80-100%

Hematopoietic:

* Granulocyte count at least 2,000/mm^3
* Platelet count at least 150,000/mm^3

Hepatic:

* Bilirubin within upper limits of normal (ULN)
* Alkaline phosphatase no greater than 1.5 times ULN
* AST no greater than 1.5 times ULN
* No chronic active hepatitis

Renal:

* Creatinine within ULN

Cardiovascular:

* No prior atrial or ventricular arrhythmias
* No history of congestive heart failure
* No myocardial infarction within the past 6 months
* No uncontrolled hypertension

Neurologic:

* No pre-existing motor or sensory neuropathy greater than grade 1

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No active infection
* No history of second malignancy except adequately treated basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* No prior endocrine therapy

Radiotherapy:

* No prior radiotherapy

Surgery:

* No prior surgery
* No prior surgical biopsy of breast nodule

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 1996-10; Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianni Bonadonna, MD, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (28):
- Kaiser Franz Josef Hospital, Vienna, Austria
- Radiotherapy Institute, Ostrava-Poruba, Czechia
- University of Tartu, Tartu, Estonia
- Frauenklinik Vom Roten Kreuz, Munich, Germany
- Hungary (2):
  - Semmelweis University, Budapest
  - Uzsoki Hospital, Budapest
- Italy (5):
  - Policlinico Monteluce, Perugia
  - Ospedale St. Santa Chiara, Pisa
  - Centro di Riferimento Oncologico - Aviano, Trento
  - Universita Degli Studi di Udine, Udine
  - Ospedale San Bortolo, Vicenza
- Latvian Cancer Center, Riga, Latvia
- Poland (4):
  - Regional Center of Oncology, Bydgoszcz
  - Jagiellonian University, Krakow (Cracow)
  - Szpital Kliniczny NR 1, Poznan
  - Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw
- Russia (5):
  - Russian Academy of Medical Sciences Cancer Research Center, Moscow
  - Moscow Clinical Dispenser, Moscow
  - N. A. Semashko Central Clinical Hospital, Moscow
  - Regional Oncology Clinic, Murmansk
  - Petrov Research Institute of Oncology, Saint Petersburg
- St. Elizabeth Cancer Institute Hospital, Bratislava, Slovakia
- Spain (6):
  - Hospital de la Santa Cruz I Sant Pau, Barcelona
  - Hospital General Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario - Malaga, Málaga
  - Instituto Valenciano De Oncologia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia

REFERENCES:
- [Result] Gianni L, Baselga J, Eiermann W, Porta VG, Semiglazov V, Lluch A, Zambetti M, Sabadell D, Raab G, Cussac AL, Bozhok A, Martinez-Agullo A, Greco M, Byakhov M, Lopez JJ, Mansutti M, Valagussa P, Bonadonna G. Phase III trial evaluating the addition of paclitaxel to doxorubicin followed by cyclophosphamide, methotrexate, and fluorouracil, as adjuvant or primary systemic therapy: European Cooperative Trial in Operable Breast Cancer. J Clin Oncol. 2009 May 20;27(15):2474-81. doi: 10.1200/JCO.2008.19.2567. Epub 2009 Mar 30. PMID 19332727